CLINICAL TRIAL: NCT06453278
Title: Validation of Diabetes Risk Assessment in Dentistry Score (DDS) in India: a Screening Tool to Identify Prediabetes and Undiagnosed Type 2 Diabetes in Dental Settings
Brief Title: (DDS) in India: a Screening Tool to Identify Prediabetes and Undiagnosed Type 2 Diabetes in Dental Settings
Status: Not yet recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: DR.ADITIPERIO
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: PreDiabetes; Type2diabetes; Periodontitis
MeSH Terms: conditions — Prediabetic State; Periodontitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study group will comprise of consenting adults aged 40 years and above.: A) INTERVIEW Demographic data, family history of type 2 diabetes mellitus and periodontal treatment history is obtained.
  BODY MASS INDEX (BMI) CALCULATION C) ORAL EXAMINATION-POCKET PROBING DEPTH (PPD) MEASUREMENT PPD Measurement of PPD will be done using a periodontal probe and mouth mirror. Measurement will be done on all teeth present in the mouth (except third molars) at six sites per tooth: mesio-buccal, mid-buccal, distobuccal, mesio-lingual, mid-lingual and distolingual.
  The number of sites with ≥5-mm probing pocket depth will be recorded on the DDS proforma. The total DDS point score will be obtained by adding all individual variable scores, ranging from 0 to 22.
  BIOCHEMICAL MEASUREMENT ( HbA1c levels in blood):
  All participants will be asked for providing blood sample for evaluation of HbA1c levels.

SUMMARY:
This study is conducted to evaluate validity of Diabetes Risk Assessment in Dentistry Score (DDS) in Indian population as a screening tool to identify patients with prediabetes and undiagnosed type 2 diabetes in dental setting. The DDS score of the patient will be correlated with the HbA1c levels and periodontal status of the patient. Such a study has been conducted in Germany but none has been validated in Indian population. Hence this study aims to assess the performance of DDS screening tool in Indian population.

DETAILED DESCRIPTION:
BACKGROUND- Most of the models for T2DM risk assessment exist for use in medical settings and include data which is commonly unavailable to dentists. To overcome the limitation of applicability of existing diabetes-risk assessment tools in dental settings, the Diabetes Risk Assessment in Dentistry Score (DDS) was developed utilizing measures routinely available to dentists. It has been developed and validated in a German population and found to perform broadly at par with those validated for use in medical settings. RATIONALE-Models developed in a specific population need to be validated in other populations before they can be adopted. The DDS screening tool has not been validated in Indian population till date. OBJECTIVES- To assess performance of DDS screening tool in predicting the risk of prediabetes and type 2 diabetes mellitus among individuals seeking dental consultation in Indian population. METHODS-The study participants will include individuals seeking dental consultation at a university teaching hospital in India. All participants will undergo DDS risk-assessment followed by measurement of serum HbA1c levels to establish diagnosis of health, prediabetes or undiagnosed T2DM. EXPECTED OUTCOMES-It is expected that the DDS screening model performs well in Indian population, with scope for incorporation of the model during regular dental visits.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria-adults aged ≥ 40 years

Exclusion Criteria:

* Individuals with existing physician-diagnosed diabetes (of any kind)
* Pregnant females

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be drawn from consecutive eligible adults attending the regular out patient department (OPD) of PGIDS, Rohtak. All individuals will be required to provide written informed consent before enrolment in the study. Inclusion criteria-adults aged ≥ 40 years Exclusion criteria-
  1. Individuals with existing physician-diagnosed diabetes (of any kind)
  2. Pregnant females
Sampling Method: Non-Probability Sample
Enrollment: 1746 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To correlate DDS score with HbA1c levels in Indian population. | 15-18 months
  Consecutive patients visiting the dental clinic will be asked to answer questions regarding symptoms of diabetes and glycemic control in an interview format. Blood samples from the patients will then be collected and Hba1c levels of the participant will be determined.
To determine prevalence of prediabetes and undiagnosed type 2 diabetes in dental patients. | 15-18 months
  Screening for risk of diabetes will be done by interviewing the patients visiting the dental out patient department. The DDS risk score for the patient will be calculated and prevalence of prediabetic and undiagnosed cases of type 2 diabetes mellitus will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: ADITI SANGWAN, MDS, Principal Investigator — Post graduate institute of Dental Sciences ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No